CLINICAL TRIAL: NCT03083314
Title: SELECTIVE AXILLARY LYMPH NODE DISSECTION VS COMPLETE AXILLARY DISSECTION: A RANDOMISED CLINICAL TRIAL TO ASSESS THE PREVENTION OF LYMPHEDEMA IN BREAST CANCER TREATMENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RF-2013-02355260
Record Dates: First submitted 2017-03-02; First posted 2017-03-20 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: The proposed study is a 2-arm (1:1 allocation) prospective randomised trial. The control arm consists of patients randomized to ALND, the study arm is patients randomized to SAD.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SELECTIVE AXILLARY LYMPH NODE DISSECTION (SAD) (Experimental)
  Interventions: Procedure: SELECTIVE AXILLARY LYMPH NODE DISSECTION (SAD)
- COMPLETE AXILLARY DISSECTION (ALND) (Active Comparator)
  Interventions: Procedure: COMPLETE AXILLARY DISSECTION (ALND)

INTERVENTIONS:
Procedure: SELECTIVE AXILLARY LYMPH NODE DISSECTION (SAD)
  Arms: SELECTIVE AXILLARY LYMPH NODE DISSECTION (SAD)
Procedure: COMPLETE AXILLARY DISSECTION (ALND)
  Arms: COMPLETE AXILLARY DISSECTION (ALND)

SUMMARY:
This is a pilot study at the National Cancer Institute (INT) of Milan evaluated the feasibility of selective axillary dissection (SAD) which preserved the lymphatic drainage of the arm. Lymph nodes draining the arm are identified following radiotracer injection and lymphoscintigraphy, a technique called axillary reverse mapping (ARM). SAD was found feasible in 75% of patients. Furthermore only 9% had BCRL after SAD compared to 33% after axillary lymph node dissection (ALND).

DETAILED DESCRIPTION:
To evaluate the efficacy, safety and cost reduction of SAD compared to standard ALND, we propose a prospective 2-arm randomised trial. The control arm consists of patients randomized to ALND, the study arm consists of patients randomized to SAD.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with operable breast cancer who are candidates for ALND, irrespective of the type of breast surgery performed or adjuvant treatments administered.
* Patients who sign the informed consent form after explanation of trial aims by a senologist involved in the study.
* Patients able to attend INT for regular follow-up as required by study protocol.

Exclusion Criteria:

* Massive axillary metastasis (N2 AJCC).
* Previous surgery to controlateral axillary region.
* Previous radiotherapy to ipsilateral or controlateral regional lymph nodes.
* Non compliance with any inclusion criterion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2014-06-12 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2020-12-04 (Actual)

PRIMARY OUTCOMES:
To compare the occurrence of breast-cancer-related lymphoedema (BCRL) after selective axillary dissection (SAD) and after axillary lymph node dissection (ALND) | 36 months
  For this purpose patients enrolled will receive a physical assessment one month after surgery, with evaluation at 6 and 12 months after surgery that includes oncological assessment, physical assessment, lymphoscintigraphy, and self-evaluation questionnaire to assess the presence BCRL.

SECONDARY OUTCOMES:
Safety of the selective axillary dissection (SAD) procedure by assessing the occurrence of axillary relapses during follow-up due to incomplete resection of axillary lymph nodes. | 36 months
  to assess the potential for residual disease in the axilla after SAD by evaluating the status, in the ALND arm, of nodes that are spared and assess the occurrence of axillary relapses during follow-up due to incomplete resection of axillary lymph nodes.

OTHER OUTCOMES:
To compare costs in the axillary lymph node dissection (ALND) and selective axillary dissection (SAD) arms | 36 months
  To compare costs in the ALND and SAD arms including: lymphoscintigraphy, time required for surgery, and treatments required for lymphedema during follow up.

CONTACTS AND LOCATIONS:
Locations (1):
- Massimiliano Gennaro, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gennaro M, Maccauro M, Sigari C, Casalini P, Bedodi L, Conti AR, Caraceni A, Bombardieri E. Selective axillary dissection after axillary reverse mapping to prevent breast-cancer-related lymphoedema. Eur J Surg Oncol. 2013 Dec;39(12):1341-5. doi: 10.1016/j.ejso.2013.09.022. Epub 2013 Oct 3. PMID 24113621
- [Result] Schunemann E Jr, Doria MT, Silvestre JB, Gasperin P Jr, Cavalcanti TC, Budel VM. Prospective study evaluating oncological safety of axillary reverse mapping. Ann Surg Oncol. 2014 Jul;21(7):2197-202. doi: 10.1245/s10434-014-3626-5. Epub 2014 Mar 6. PMID 24599413
- [Result] Agresti R, Martelli G, Sandri M, Tagliabue E, Carcangiu ML, Maugeri I, Pellitteri C, Ferraris C, Capri G, Moliterni A, Bianchi G, Mariani G, Trecate G, Lozza L, Langer M, Rampa M, Gennaro M, Greco M, Menard S, Pierotti MA. Axillary lymph node dissection versus no dissection in patients with T1N0 breast cancer: a randomized clinical trial (INT09/98). Cancer. 2014 Mar 15;120(6):885-93. doi: 10.1002/cncr.28499. Epub 2013 Dec 5. PMID 24323615
- [Result] Giuliano AE, Hunt KK, Ballman KV, Beitsch PD, Whitworth PW, Blumencranz PW, Leitch AM, Saha S, McCall LM, Morrow M. Axillary dissection vs no axillary dissection in women with invasive breast cancer and sentinel node metastasis: a randomized clinical trial. JAMA. 2011 Feb 9;305(6):569-75. doi: 10.1001/jama.2011.90. PMID 21304082
- [Result] Shah C, Wilkinson JB, Baschnagel A, Ghilezan M, Riutta J, Dekhne N, Balaraman S, Mitchell C, Wallace M, Vicini F. Factors associated with the development of breast cancer-related lymphedema after whole-breast irradiation. Int J Radiat Oncol Biol Phys. 2012 Jul 15;83(4):1095-100. doi: 10.1016/j.ijrobp.2011.09.058. Epub 2011 Nov 16. PMID 22099041
- [Result] Ozcinar B, Guler SA, Kocaman N, Ozkan M, Gulluoglu BM, Ozmen V. Breast cancer related lymphedema in patients with different loco-regional treatments. Breast. 2012 Jun;21(3):361-5. doi: 10.1016/j.breast.2012.03.002. Epub 2012 Mar 27. PMID 22460058
- [Result] Cheville A. Prevention of lymphoedema after axillary surgery for breast cancer. BMJ. 2010 Jan 12;340:b5235. doi: 10.1136/bmj.b5235. No abstract available. PMID 20068254